CLINICAL TRIAL: NCT05985395
Title: An Intervention to Promote Exercise in Adults With Heart Failure With Preserved Ejection Fraction
Brief Title: HEART Camp Connect: A Feasibility Study
Status: Terminated | Phase: Not Applicable | Type: Interventional
Why Stopped: R01 grant received, had to terminate preliminary research
Sponsor: University of Nebraska (Other)
Responsible Party: Sponsor
Allocation: Randomized | Model: Single Group | Masking: Single | Purpose: Health Services Research
Other Study IDs: 0914-21-FB
Record Dates: First submitted 2023-08-02; First posted 2023-08-14 (Actual); Results first posted 2025-03-20 (Actual); Last update posted 2025-12-11 (Actual); Status verified 2025-03

CONDITIONS: Heart Failure With Preserved Ejection Fraction
Keywords: exercise training; adherence; coaching

STUDY DESIGN:
Who Masked: Outcomes Assessor
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- HEART Camp Connect (Experimental): Participants will have access to a virtual exercise platform or membership to a medical exercise facility. Participants will meet with a virtual exercise coach via Zoom on a weekly basis.
  Interventions: Behavioral: HEART Camp Connect
- Usual Care (No Intervention): Participants will have access to a virtual exercise platform or membership to a medical exercise facility.

INTERVENTIONS:
Behavioral: HEART Camp Connect — Once eligible and enrolled, participants will complete 150 minutes of moderate-intensity exercise a week with help of a virtual exercise coach.
  Arms: HEART Camp Connect

SUMMARY:
This study builds on the tested and refined HEART Camp intervention which has been shown to improve long-term adherence to exercise in individuals diagnosed with heart failure. HEART Camp Connect enhances HEART Camp by delivering the coaching via videoconference and providing access to hospital-based exercise facilities and online exercise programming. This prospective study uses a 2-group, randomized repeated measures experimental design with 3 data collection points baseline, Month 3, and Month 6.

DETAILED DESCRIPTION:
Potential participants will be approached at a Heart Failure clinic at an academic medical center. As a secondary recruitment strategy, we will use a database that identifies patients who previously indicated their willingness to be contacted for clinical research.

Study personnel will obtain informed consent in person in a private room or over the phone facilitated by the academic medical center electronic consent process. Once consented, participants will complete cardiopulmonary exercise testing (CPET) to guide individual exercise prescriptions and protect against risks associated with exercise. CPET results that preclude safe exercise training (arrhythmia) or those with CPET results indicating cardio-respiratory fitness (females with maximum oxygen consumption ≥ 21ml/kg/min and males with oxygen consumption ≥ 24 ml/kg/min) will be withdrawn from the study.

Participants will be given instruction on the use of the heart rate monitor. Participants will wear their monitor exercise sessions for heart rate monitoring. Participants will also receive educational training via videos on topics such as exercising with heart failure, how medications impact exercise, and nutrition.

Participants will be instructed to wear a heart rate monitor and strive to meet a goal of 150 minutes of moderate-intensity exercise per week. Minutes toward adherence goals for the study will be calculated as time spent participating in a moderate-intensity activity and determined by their CPET results and personalized exercise prescription.

Each participant will be given access to an Omaha-based exercise coach that he/she will meet with weekly over Zoom for 30 minutes. Coaches will discuss exercise over the past week including problems, issues, concerns. Goals will be set, reviewed, assessed, and revised each week. For virtual exercise, all participants will access a Virtual Wellness Center.

ELIGIBILITY:
Inclusion Criteria:

* Diagnosis of heart failure (HF) with an ejection fraction (EF) ≥50%
* Age ≥18 years
* English-speaking
* Echocardiogram in prior 12 months
* Stable pharmacologic therapy in past 30 days

Exclusion Criteria:

* Score<6 on a diagnostic algorithm
* Life-limiting illness precluding study completion
* Clinical evidence of decompensated HF
* Unstable angina or marked shortness of breath on exertion at <2 metabolic equivalents
* Myocardial infarction, coronary artery bypass surgery, or biventricular pacemaker <6 weeks
* Orthopedic or neuromuscular disorders preventing participation in aerobic exercise
* Cardiopulmonary exercise test results that preclude safe exercise
* Unwilling/unable to complete pre-randomization procedures
* Pregnancy
* Implantable cardioverter-defibrillator

Min Age: 18 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Enrollment: 11 (Actual)
Dates: Start 2022-03-28 (Actual); Primary Completion 2023-11-20 (Actual); Study Completion 2023-11-20 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Windy W Alonso, PhD, RN, Principal Investigator — University of Nebraska
Locations (1):
- University of Nebraska Medical Center, Omaha, Nebraska, United States

IPD SHARING:
Plan to Share IPD: No

RESULTS

PARTICIPANT FLOW:
Period: Overall Study
Arm/Group | HEART Camp Connect | Usual Care
Started | 7 | 4
Completed | 4 | 3
Not Completed | 3 | 1
Not completed — Physician Decision | 2 | 1
Not completed — Withdrawal by Subject | 1 | 0

BASELINE CHARACTERISTICS:
Groups:
- Total: Total of all reporting groups
Arm/Group | HEART Camp Connect | Usual Care | Total
Number analyzed (Participants) | 4 | 3 | 7
Age, Continuous [Mean (Standard Deviation); unit: years] | 69.5 (14.01) | 70.3 (6.4) | 69.9 (10.6)
Sex: Female, Male [Count of Participants; unit: Participants] — As reported in medical record
  Participants
    Female | 3 | 3 | 6
    Male | 1 | 0 | 1
Race (NIH/OMB) [Count of Participants; unit: Participants]
  American Indian or Alaska Native | 0 | 0 | 0
  Asian | 0 | 0 | 0
  Native Hawaiian or Other Pacific Islander | 0 | 0 | 0
  Black or African American | 0 | 1 | 1
  White | 4 | 2 | 6
  More than one race | 0 | 0 | 0
  Unknown or Not Reported | 0 | 0 | 0
Region of Enrollment [Number; unit: participants]
  United States | 4 | 3 | 7
Exercise Adherence [Count of Participants; unit: Participants] — At baseline all participants were sedentary and not participating in exercise
  Participants | 0 | 0 | 0
Kansas City Cardiomyopathy Questionnaire Overall Summary Score [Mean (Standard Deviation); unit: units on a scale] | 46.3 (16.3) | 48.7 (17.1) | 47.7 (15.4)

OUTCOME MEASURES:

1. Primary Outcome: Exercise Adherence
Description: Exercise adherence is defined as a count of the number of participants meeting 120 minutes or more of moderate intensity exercise per week at the prespecified time point of 3 months.
Time Frame: 3 months
Measure: Count of Participants; unit: Participants
Arm/Group | HEART Camp Connect | Usual Care
Number analyzed (Participants) | 4 | 3
Participants | 1 | 1

2. Secondary Outcome: Kansas City Cardiomyopathy Questionnaire (KCCQ) Overall Summary Score
Description: KCCQ measures heart failure related health status. The overall summary score ranges from 0 to 100, with higher scores indicating better health status, typically interpreted in 25-point ranges as: very poor to poor (0-24), poor to fair (25-49), fair to good (50-74), and good to excellent (75-100). A change in score of 5 points or more is considered clinically meaningful.
Time Frame: 3 months
Population: 1 participant in the intervention group was missing KCCQ data for 3 months
Measure: Mean (Standard Deviation); unit: units on a scale
Arm/Group | HEART Camp Connect | Usual Care
Number analyzed (Participants) | 3 | 3
units on a scale | 56.7 (14.3) | 57.4 (16.1)

3. Other Pre Specified Outcome: Smart Devices
Description: Measures is a count of the number of potential participants without smart devices at baseline. Participants without a smart device are loaned one for the duration of the study.
Time Frame: Baseline
Measure: Count of Participants; unit: Participants
Arm/Group | HEART Camp Connect | Usual Care
Number analyzed (Participants) | 4 | 3
Participants | 2 | 1

ADVERSE EVENTS:
Time Frame: Events data collected for 3 months
Description: We used standard definitions.
Arm/Group | HEART Camp Connect | Usual Care
All-Cause Mortality (participants affected / at risk) | 0/4 | 0/3
Serious Adverse Events (participants affected / at risk) | 0/4 | 0/3
Other Adverse Events (participants affected / at risk) | 0/4 | 0/3

LIMITATIONS AND CAVEATS:
We initially planned to enroll 25 participants per arm but upon receipt of R01 funding the funds for this pilot study had to be forfeited. Therefore, only 7 were enrolled and completed. Data collection and analyses were limited.

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: Yes; Agreement restricts PI disclosure of results: No

DOCUMENTS (2):
  • Study Protocol and Statistical Analysis Plan (2023-12-26): https://cdn.clinicaltrials.gov/large-docs/95/NCT05985395/Prot_SAP_000.pdf
  • Informed Consent Form (2024-11-13): https://cdn.clinicaltrials.gov/large-docs/95/NCT05985395/ICF_001.pdf